CLINICAL TRIAL: NCT01287845
Title: Open-label, Multi Center PET/CT Study for Investigation of Safety, Tolerability, Biodistribution and Diagnostic Performance of the 18F Labeled PET Tracer BAY1075553 Following a Single Intravenous Administration of 300 MBq in Patients With Prostate Cancer as Well as Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Tolerability of the Tracer in PET/CT in Healthy Volunteers.
Brief Title: PET/CT (Positron Emission Tomography/Computed Tomography) Imaging for Safety and Tolerability and Diagnostic Performance of BAY1075553 in Patients With Prostate Cancer and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15117; 2010-022031-11 (EudraCT Number)
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Diagnostic Imaging
Keywords: Prostate cancer; Neoplasm; Diagnostic Imaging; PET (Positron Emission Tomography) -tracer; PET-diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY1075553
- Arm 2 (Experimental)
  Interventions: Drug: BAY1075553

INTERVENTIONS:
Drug: BAY1075553 — Cancer patients, single intravenous bolus injection of 300 MBq BAY1075553 over 60 seconds on the treatment day 1
  Arms: Arm 1
Drug: BAY1075553 — Healthy volunteers for dosimetry, single intravenous bolus injection of 300 MBq BAY1075553 over 60 seconds on the treatment day 1
  Arms: Arm 2

SUMMARY:
PET/CT imaging study for evaluation of safety and tolerability and diagnostic performance of BAY1075553 in patients with prostate cancer and in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Healthy volunteers only

  -- Males ≥ 40 years of age
* Part 2: Prostate cancer patients

  * Males ≥ 18 years of age
  * Serum PSA (Prostate-Specific Antigen) value above normal.
  * Patients had an MRI and/or a positive [11C] - or [18F] -choline PET/CT for primary diagnosis (Note: MRI and [11C]-or [18F]-choline PET/CT are optional for primary prostate cancer patients) or recurrence detection of prostate cancer and the primary cancer disease (adenocarcinoma) is histologically confirmed
  * Patients with primary prostate cancer have to be scheduled for prostatectomy
  * In patients with primary prostate cancer, histopathological evaluation has to show an adenocarcinoma with a Gleason score of 3 + 3 or higher in at least two biopsies at any location in the prostate
  * Patients with advanced primary or recurrent prostate cancer and a high likelihood to display lymph node metastasis, ideally scheduled for explorative pelvic lymphadenectomy, are to be preferably included
* Part 3: Prostate cancer patients -- The criteria for eligibility of part 3 are identical to the ones of part 2. Except it is now no longer a preference but mandatory to only enrol patients with a presumably high likelihood of metastatic disease, especially lymph node metastasis.

Exclusion Criteria:

* Concurrent severe and/or uncontrolled and/or unstable medical disease other than prostate cancer (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY1075553, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
* Acute renal insufficiency of any intensity, either due to hepato-renal syndrome or occurring in the peri-operative liver transplantation period
* Active inflammatory bowel disease within the last 6 months
* Acute prostatitis requiring medical treatment within the last 6 months
* A non-urologic bacterial infection requiring active treatment with antibiotics within 3 months
* Active other malignancy (except basal cell or squamous cell skin cancer) within the last 2 years
* Patients with primary prostate cancer only: androgen ablation within 3 months before planned treatment
* Subject fulfils criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety parameters, for example laboratory and electrocardiogram abnormalities | Day 2
Effective radiation dose given in mSv (milliSievert) in healthy volunteers | Day 1

SECONDARY OUTCOMES:
Overall lesion detection rate | Day 1
Lesion detection rate in comparison to histology, where available (cancer lesion detection rate) | Day 1
Lesion detection rate in comparison to MRI (Magnetic Resonance Imaging) and/or [11C] (11Carbon)- or [18F] (18Fluor)-choline PET/CT (whenever available) | Day 1
Accumulation score in all lesions identified with BAY1075553 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Ann Arbor, Michigan, United States
- Linz, Austria